CLINICAL TRIAL: NCT04071119
Title: The Neural Mechanisms Associated With Alcohol and Cigarette Craving in Alcohol Use Disorder Smokers During Oxytocin Treatment
Brief Title: Alcohol and Cigarette Craving During Oxytocin Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Kimberly Goodyear, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 22301; K01AA026874 (NIH)
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Use Disorder; Smoking
Keywords: oxytocin; craving; alcohol use disorder; smoking; cigarettes; drinking; functional magnetic resonance imaging; cue-reactivity
MeSH Terms: conditions — Alcoholism; Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin nasal spray (Active Comparator)
  Interventions: Drug: Oxytocin nasal spray
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — Participants administer the oxytocin (40 IU) twice a day for 5 - 7 days
  Arms: Oxytocin nasal spray
Drug: Placebo — Participants administer the placebo (40 IU) twice a day for 5 - 7 days
  Arms: Placebo

SUMMARY:
This proposed research seeks to examine the behavioral and neural substrates of intranasal oxytocin compared to placebo on alcohol cue-induced alcohol and cigarette craving smokers with an alcohol use disorder (AUD). Non treatment-seeking smokers with an AUD will be recruited to participate in a between-subjects, placebo-controlled, randomized pilot functional magnetic resonance imaging (fMRI) study. Participants will undergo an fMRI scan in conjunction with an alcohol-olfactory cue-reactivity task. Secondary assessments will include alcohol and cigarette craving, alcohol and cigarette consumption, physiological measures (heart rate and blood pressure) and mood measures.

ELIGIBILITY:
Inclusion Criteria:

1. male or female
2. 18 to 55 years of age
3. meet criteria for Alcohol Use Disorder DSM-5 diagnosis
4. meet the National Institute on Alcohol Abuse and Alcoholism criteria for heavy-drinking
5. smoke at least ≥5 cigarettes/day for at least a year, verified with breath carbon monoxide level > 5 ppm
6. in good health as confirmed by medical history, physical examination and lab tests
7. willing to take the medication and adhere to the study procedures
8. breath alcohol concentration (BrAC) = 0.00 at each visit
9. understand informed consent and questionnaires written in English at an 8th grade level
10. right-handedness
11. normal to normal-corrected vision

Exclusion Criteria:

1. positive urine test for pregnancy
2. women who are breast-feeding
3. body mass index > 40
4. current or prior history of any clinically significant disease, cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders, positive hepatitis or HIV test that could affect study participation, as determined by the study physician
5. history of suicide attempts
6. current diagnosis of substance dependence other than alcohol, nicotine or cannabis as assessed by self-report and urine toxicology screen at baseline
7. current use of psychoactive medications or any medication that may interact with oxytocin
8. history of hypersensitivity to oxytocin
9. chronic rhinitis or sinusitis
10. clinically significant electrolyte abnormalities
11. vasoconstricting medications or prostaglandins
12. clinically significant medical abnormalities: unstable hypertension, bilirubin >150% of the upper normal limit (UNL), ALT/AST >500% the UNL, creatinine clearance ≤60 dl/min)
13. significant alcohol withdrawal symptoms, defined as a CIWA-Ar > 8
14. positive urine drug screen at baseline for any excluded substances
15. individuals seeking treatment
16. meets DSM-5 criteria for a diagnosis of schizophrenia, bipolar disorder, or other psychoses
17. claustrophobia
18. any contraindications with the MRI machine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Alcohol craving | 1 day
  average alcohol craving during the cue-reactivity task
Cigarette craving | 1 day
  average cigarette craving during the cue-reactivity task
Brain activity | 1 day
  BOLD response when comparing alcohol to neutral cues during fMRI

SECONDARY OUTCOMES:
Alcohol and cigarette consumption | 5-7 days
  alcohol and cigarette consumption assessed by the Timeline Followback

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No